CLINICAL TRIAL: NCT03327701
Title: The Effect of Benralizumab on Lung Physiology, Exercise-induced Bronchoconstriction and General Health Status: an Exploratory Mechanistic Study
Brief Title: The Effect of Benralizumab on Exercise-induced Bronchoconstriction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Louis-Philippe Boulet (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Louis-Philippe Boulet, MD FRCPC FCCP, Respirologist, Laval University
Organization: Laval University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CER-21525
Record Dates: First submitted 2017-10-19; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Asthma, Exercise-Induced
Keywords: Exercise-induced bronchoconstriction; Benralizumab; Antiinterleukin 5 receptor α monoclonal antibody
MeSH Terms: conditions — Asthma, Exercise-Induced | interventions — benralizumab

STUDY DESIGN:
Intervention Model Description: This study is a parallel study, double-blind, placebo controlled randomized trial, with a ratio placebo-active drug 1:2.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study will be conducted under double-blind conditions. Neither the subject nor the investigator and clinical site personnel will know which medication is administered. The medication given will be determined according to a randomization table handled by a collaborating IUCPQ-UL pharmacist. Only the pharmacist responsible for preparing the medication for the randomized patients will have access to information on treatment allocations (unblended). Benralizumab and placebo solutions for injection in an accessorized pre-filled syringe (PFS) will have the same packaging.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Active Comparator): Subjects will receive benralizumab 30 mg (subcutaneous) every 4 weeks for three doses followed by a fourth dose 8 weeks later.
  Interventions: Drug: Benralizumab
- Placebo (Placebo Comparator): Subjects will receive placebo 30 mg (subcutaneous) every 4 weeks for three doses followed by a fourth dose 8 weeks later.
  Interventions: Drug: Benralizumab

INTERVENTIONS:
Drug: Benralizumab — Subjects will receive benralizumab 30 mg (subcutaneous) every 4 weeks for three doses followed by a fourth dose 8 weeks later.

SUMMARY:
Severe asthma affects 5-10% of more than 300 million asthmatics. Ten to twenty percent of individuals suffering from asthma do not respond well to current treatment due to the complexity of the different mechanisms underlying asthma pathogenesis, and sometimes due to an insufficient effect of treatment on underlying airway inflammation. Consequently, some asthmatics have poorer quality of life due to: frequent asthma symptoms, regular medical or emergency visits, limitation in their activities of daily living, including exercise. It is believed that the benralizumab can help to reduce airway inflammation and thus improve exercise tolerance in individuals with asthma. The main objective of this study is to determine the effect of benralizumab on exercise-induced bronchoconstriction (EIB) and exercise tolerance in moderate to severe eosinophilic asthmatics, in comparison with baseline values and a placebo treatment.

DETAILED DESCRIPTION:
Subjects will receive benralizumab every 4 weeks for three doses followed by a fourth dose 8 weeks later. On baseline and after 4, 16 and 20 weeks, subjects will be assess for airway responsiveness to exercise and exercise tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for study participants must be obtained prior to any study related procedures being performed and according to local guidelines;
2. Asthma diagnosis according to current guidelines;
3. General good health as declared by the investigator;
4. Respiratory symptoms such as wheeze, shortness of breath, chest tightness or cough during physical activity;
5. Moderate to severe eosinophilic asthma (Inhaled corticosteroids, 250 mcg/day fluticasone equivalent or more and long acting beta2-agonists, stable for at least one month);
6. Sufficient adherence to maintenance therapy (from questionnaire and pharmacy reports: adherence to at least 80% of medication prescribed on both);
7. Baseline blood eosinophil counts of at least 300 cells/ul and/or sputum eosinophil of at least 3%;
8. Exercise less than 4 hours per week and remain stable through the study;
9. Presence of EIB: A post-exercise fall in FEV1 of at least 10% from baseline;
10. Pre-bronchodilator FEV1 at screening of at least 70% of the predicted value;
11. Women of childbearing potential (WOCBP) must use an effective form of birth control (confirmed by the investigator). Effective forms of birth control include: true sexual abstinence, a vasectomized sexual partner, Implanon, female sterilization by tubal occlusion, any effective intrauterine device/levonorgestrel Intrauterine system, Depo-Provera™ injections, oral contraceptive, and Evra Patch™ or Nuvaring™. WOCBP must agree to use effective method of birth control, as defined above, from enrolment, throughout the study duration and 20 weeks after last dose of study product, and have negative serum pregnancy test result on Visit 1;

    a. Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrheic for 12 months prior to the planned date of randomization without an alternative medical cause. The following age-specific requirements apply:
12. Women <50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment. They also need follicle stimulating hormone (FSH) levels in the postmenopausal range.
13. Women ≥50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.

Exclusion Criteria:

1. Respiratory tract infection within 6 weeks preceding enrolment;
2. Asthma exacerbation in the last month;
3. Use of prednisone in the last 30 days;
4. Current lung disease other than moderate to severe eosinophilic asthma;
5. History of clinically significant hypotensive episodes or symptoms of fainting, dizziness, or light headedness, as judged by the investigator;
6. Any history or symptoms of uncontrolled cardiovascular disease, particularly coronary artery disease, arrhythmias, hypertension, or congestive heart failure;
7. Any history or symptoms of significant neurologic disease, including transient ischemic attack (TIA), stroke, seizure disorder, or behavioural disturbances;
8. Any history or symptoms of clinically significant autoimmune disease;
9. Any history of clinically significant haematologic abnormality, including coagulopathy or any history of chronic treatment with anti-coagulants (e.g. warfarin, etc.) or anti-platelet agent (e.g. aspirin, etc.);
10. Clinically significant abnormalities in laboratory test results at enrolment and during the screening period (including complete blood count, coagulation, chemistry panel and urinalysis) unless judged not significant by the investigator;
11. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥2.5 times the upper limit of normal (ULN) confirmed during screening period;
12. Being pregnant or lactating or have positive serum pregnancy test at enrolment or positive urine pregnancy test during the study;
13. Use of nonsteroidal anti-inflammatory drugs (NSAIDs) 72 hours before or aspirin prn within 7 days of enrolment (Visit 1), as judged by the investigator;
14. Current smokers. Ex-smokers must not have smoked for a minimum of 12 months, and should not have a smoking history ≥10 pack years. Subjects who administer nicotine in other forms (patches, chew tobacco, etc.) will also be excluded from the study;
15. Concomitant disease or condition which could interfere with the conduct of the study, or for which the treatment might interfere with the conduct of the study, or which would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study, including, but not limited to, cancer, alcoholism, drug dependency or abuse, or psychiatric disease;
16. History of cancer in last 5 years:
17. Alcohol or drug abuse (past or present);
18. Subject who is scheduled to be admitted to hospital or undergo in-subject surgery during the study;
19. History of anaphylaxis to any biologic therapy or vaccine;
20. History of Guillain-Barré syndrome;
21. A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with, or has failed to respond to standard of care therapy;
22. Positive hepatitis B surface antigen, or hepatitis C virus antibody serology, or a positive medical history for hepatitis B or C. Subjects with a history of hepatitis B vaccination without history of hepatitis B are allowed to enrol;
23. A history of known immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test;
24. Use of immunosuppressive medication (including but not limited to: methotrexate, troleandomycin, cyclosporine, azathioprine, intramuscular long-acting depot corticosteroid, oral corticosteroid, or any experimental anti-inflammatory therapy) within 3 months prior to the date informed consent is obtained;
25. Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent is obtained;
26. Receipt of any marketed (e.g. omalizumab) or investigational biologic within 4 months or 5 half-lives prior to randomization is obtained, whichever is longer;
27. Receipt of live attenuated vaccines 30 days prior to the date of randomization

    - Receipt of inactive/killed vaccinations (e.g., inactive influenza) are allowed provided they are not administered within 1 week before/after any IP administration.
28. Previously received benralizumab (MEDI-563);
29. AstraZeneca staff involved in planning and/or conducting the study;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change in post-exercise fall in expiratory flows | Baseline and after 4, 16 and 20 weeks
  Maximal fall in forced expiratory volume in one second (FEV1) post-exercise challenge

SECONDARY OUTCOMES:
Change in exercise tolerance | Baseline and after 4, 16 and 20 weeks
  Endurance time on a steady-state exercise

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval

IPD SHARING:
Plan to Share IPD: No